CLINICAL TRIAL: NCT04132271
Title: Effect of Swallowing Rehabilitation Complemented With Nutritional Treatment on the Nutritional Status of Oropharyngeal Dysphagia Patients
Brief Title: Swallowing and Nutritional Treatment on OD Patients
Acronym: OD
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Hospital General de Mexico (Other Government)
Responsible Party: Principal Investigator, Nallely Bueno Hernández, Investigator In Medical Science B, Hospital General de Mexico
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: DI/19/301/03/003
Record Dates: First submitted 2019-10-08; First posted 2019-10-18 (Actual); Last update posted 2019-10-18 (Actual); Status verified 2019-10

CONDITIONS: Oropharyngeal Dysphagia
Keywords: oropharyngeal, dysphagia, nutrition
MeSH Terms: conditions — Deglutition Disorders

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Personalized diet (Experimental): Personalized diet during the swallowing rehabilitation
  Interventions: Other: Personalized diet
- Control (Active Comparator): Nutritional recommendations during the swallowing rehabilitation
  Interventions: Other: Control

INTERVENTIONS:
Other: Personalized diet — Modified texture and volumen diet according to the OD specifications
  Arms: Personalized diet
Other: Control — Nutritional Recommendations according to the OD specifications
  Other Names: Nutritional Recommendations
  Arms: Control

SUMMARY:
Dysphagia is a difficulty during the swallowing process (transportation food from the mouth to the stomach. Oropharyngeal Dysphagia (OD) is diagnosed by videofluoroscopy and faringolaringoscopy. OD threatens the efficacy and safety of swallowing, contributing to an increased risk of aspiration and pneumonia. There are different interventions aimed to change and improve the physiology of swallowing; however, OD can be an important predictor of the progression of malnutrition in different types of patients. Malnutrition is defined as an acute or chronic disease whereby an energy imbalance, lack of energy, protein or other nutrients causes measurable and adverse effects on body composition, functional and clinical outcomes. In addition, it leads to a decrease in the quality of life.

Objective: To establish a strategy of nutritional treatment and swallowing rehabilitation in patients with dysphagia.

Hypothesis: An adequate nutritional intervention in content and consistency, combined with swallowing rehabilitation in patients with dysphagia, will improve the nutritional status and clinical evolution of patients with dysphagia.

DETAILED DESCRIPTION:
Introduction: Dysphagia is a difficulty during the swallowing process (transportation food from the mouth to the stomach. Oropharyngeal Dysphagia (OD) is diagnosed by videoflouroscopy and faringolaringoscopy and it is frequently associated with neurodegenerative problems. OD threatens the efficacy and safety of swallowing, contributing to an increased risk of aspiration and pneumonia.

Problem statement: There are different interventions aimed to change and improve the physiology of swallowing; however, OD can be an important predictor of the progression of malnutrition in different types of patients. Malnutrition is defined as an acute or chronic disease whereby an energy imbalance, lack of energy, protein or other nutrients causes measurable and adverse effects on body composition, functional and clinical outcomes. In addition, it leads to a decrease in the quality of life.

Justification: It is essential to provide adequate nutritional interventions according to the specifications of the dysphagia in order to improve the nutritional status of these patients, as well to provide adequate early nutritional treatment when changing from tube to oral feeding, focusing on dietary factors that can significantly improve nutrition of the patient. However, there are no studies that evaluate the specific requirements for the nutritional treatment of these patients. By implementing a diet based on improving the safety and efficacy of swallowing in patients with OD, specific nutritional recommendations that impact on the rate of malnutrition and mortality of the different pathologies that present this condition could be established.

Objective: To establish a strategy of nutritional treatment and swallowing rehabilitation in patients with dysphagia.

Hypothesis: An adequate nutritional intervention in content and consistency, combined with swallowing rehabilitation in patients with dysphagia, will improve the nutritional status and clinical evolution of patients with dysphagia.

Methodology: This is a prospective randomized controlled clinical trial, in which OD patients will be recruited to participate. The participants will be receiving swallowing rehabilitation by a specialist phoniatrician. They will be randomise assigned to a special nutritional treatment during 12 weeks. Swallowing rehabilitation, laboratory analyses, anthropometric measurements and consume and quality of life questionaries will be carried out.

ELIGIBILITY:
Inclusion Criteria:

* Both sexes
* 18 to 75 years old
* Diagnosis of dysphagia
* Full phonological assessment
* Any federative entity in the country

Exclusion Criteria:

* Patients with any nephropathy
* HIV diagnosis
* Thyroid dysfunction dignosis
* Gastrostomy feeded patients
* Patients on chemotherapy
* Psychogenic Dysphagia

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 68 (Estimated)
Dates: Start 2019-12-03 (Estimated); Primary Completion 2020-02-01 (Estimated); Study Completion 2020-12-30 (Estimated)

PRIMARY OUTCOMES:
Nutritional intervention and swallowing rehabilitation on nutritional status of OD patients | Participants will be evaluated at weeks 1, 6 and 12
  Changes from baseline anthropometric, biochemical, and body composition values, at 12 weeks of nutritional intervention in OD patients

SECONDARY OUTCOMES:
Swallowing capacity | Participants will be evaluated at weeks 1, 6 and 12
  Changes from baseline of the presence or absence of food remains in the larynx and aspiration during the Fibroendoscopic Evaluation of Swallowing at 12 weeks of nutritional intervention in OD patients
Body composition analysis | Participants will be evaluated at weeks 1, 6 and 12
  Changes from baseline of the percentage of body fat, muscle and water at 12 weeks of nutritional intervention, using RJL System IV
Quality of life | Participants will be evaluated at weeks 1, 6 and 12
  Changes from baseline of WHOQOL- BREF questionary score (the higher score, the higher quality of life represents) at 12 weeks of nutritional intervention in OD patients
Anthropometric measurements | Participants will be evaluated at weeks 1, 6 and 12
  Changes from baseline of arm, waist and hips circumferences in centimeters at 12 weeks of nutritional intervention in OD patients
Nutritional Risk | Participants will be evaluated at weeks 1, 6 and 12
  Changes from baseline of malnutrition risk during the Malnutrition Universal Screening Tool score (0 = low risk; 1= medium risk 2= high risk) at 12 weeks of nutritional intervention in OD patients.
Gastrointestinal symptoms | Participants will be evaluated at weeks 1, 6 and 12
  Changes from baseline in the presence or absence of gastrointestinal symptoms according to the ROME III criteria at 12 weeks of nutritional intervention in OD patients
Dietary intake | Participants will be evaluated at weeks 1, 6 and 12
  Changes from baseline of grams of macronutrients (carbohydrates, lipids and protein) consumed, according to the 24 hours record at 12 weeks of nutritional intervention in OD patients
Blood quemistry | Participants will be evaluated at weeks 1 and 12
  Changes from baseline glucose, creatinine, high density lipoproteins, low density lipoproteins, cholesterol levels (mg/dL) at 12 weeks of nutritional intervention in OD patients
Blood chemistry | Participants will be evaluated at weeks 1 and 12
  Changes from baseline calcium, albumin, hemoglobin levels (g/dL) and iron (ug/dL) levels at 12 weeks of nutritional intervention in OD patients
Electrolytes blood levels | Participants will be evaluated at weeks 1 and 12
  Changes from baseline sodium and potasium levels (meq/L) at 12 weeks of nutritional intervention in OD patients

CONTACTS AND LOCATIONS:
Locations (1):
- Nallely Bueno Hernandez, Mexico City, Cuauhtemoc, Mexico